CLINICAL TRIAL: NCT03768128
Title: A Prospective, Multicenter Post-Market Clinical Follow-up Study to Evaluate the Safety and Performance of the Journey™ II UNI Unicompartmental Knee System
Brief Title: Safety and Performance of the Journey™ II UNI Unicompartmental Knee System
Acronym: JII-Uni
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-4049-12
Record Dates: First submitted 2018-11-27; First posted 2018-12-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-09

CONDITIONS: Non-inflammatory Degenerative Joint Disease (NIDJD) of the Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Journey™ II UNI Unicompartmental Knee System — Journey™ II UNI UKS is a CE Marked medical device. The device has been designed to treat both medial and lateral unicompartmental disease.
  It is a comprehensive system designed to allow surgeons to perform UKA. It is comprised of the following anatomic components: Oxidized zirconium femoral components Titanium tibial components with a grit-blasted surface Polyethylene tibial insert components The device is asymmetric and is available in oxidized zirconium to reduce wear and increase implant longevity.

SUMMARY:
This clinical study will evaluate the early to midterm safety and performance of the JOURNEY™ II UNI UKS in patients with non-inflammatory degenerative joint disease of the knee requiring lateral or medial knee compartment replacement. Clinical, radiographic, health economic and safety outcomes will be evaluated.

DETAILED DESCRIPTION:
To assess the safety and performance of the JOURNEY™ II UNI UKS in patients with unicompartmental degeneration of the knee by demonstrating non-inferiority of the cumulative percent implant survival in subjects with the JOURNEY™ II UNI UKS implanted, compared to a literature reference rate of 91.7% (AOA annual report 2015)12 at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria for inclusion in the study.

  1. Unicompartmental, NIDJD, including OA, traumatic arthritis, or avascular necrosis.
  2. Eighteen (18) years of age or older at the time of surgery.
  3. Skeletally mature in the judgement of the PI.
  4. Has met an acceptable preoperative medical clearance and is free of (or acceptably managed) cardiac, pulmonary, hematological, infection, or other conditions that would pose an excessive operative risk.
  5. Willing and able to participate in required follow-up visits at the investigational site and to complete study procedures and questionnaires.
  6. Consented to participate in the study by signing the EC-approved ICF.

     Exclusion Criteria:
* Subjects meeting any of the following criteria must be excluded from participation in the study.

  1. Correction of functional deformity.
  2. Revision procedures where other treatments or devices have failed.
  3. Treatment of fractures that are unmanageable using other techniques.
  4. Inadequate bone stock to support the device which would make the procedure unjustifiable, including but not limited to severe osteopenia/osteoporosis or family history of severe osteoporosis/osteopenia.
  5. Body Mass Index (BMI) > 40.
  6. Collateral ligament insufficiency.
  7. Active infection, treated or untreated, systemic or at the site of the planned surgery or previous intra-articular infections.
  8. Incomplete or deficient soft tissue surrounding the knee.
  9. Conditions that may interfere with the UKA survival or outcome, including but not limited to Paget's disease, Charcot disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, renal insufficiency or neuromuscular disease.
  10. Diagnosis of an immunosuppressive disorder.
  11. Known allergy to study device or one or more of its components.
  12. Pregnant or planning to become pregnant during the course of the study.
  13. Subject, in the opinion of the PI, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: JOURNEY™ II UNI Unicompartmental Knee System (UKS) in patients with non-inflammatory degenerative joint disease (NIDJD) of the knee requiring either medial or lateral compartment knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Implant survival 5 years postoperatively | 5 years

SECONDARY OUTCOMES:
Device-related adverse events | 5 year
  All AEs will be collected and reported
Radiographic assessments | 5 year
  To assess changes in implant fixation and bone integrity, an evaluation will be performed based upon comparison of Antero posterior and Lateral radiographs over multiple time-points. Radiographs will be also evaluated for radiolucencies, osteolysis, implant positioning, implant migration, implant loosening, periprosthetic fracture, wear of the articulating surfaces of replacement components

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - OrthoIllinois, LTD, Rockford, Illinois
- Italy (2):
  - Poliambulanza Institute Hospital Foundation, Brescia
  - Istituto Clinico Villa Aprica, Como
- Poland (2):
  - Zeromski Hospital, Krakow
  - Hospital Miejski Zabrze, Zabrze

IPD SHARING:
Plan to Share IPD: No